CLINICAL TRIAL: NCT03843762
Title: Harnessing Sleep/Circadian Rhythm Data as a Biomarker to Mitigate Health Risks
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00101670
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-02

CONDITIONS: Adolescent Behavior
Keywords: Adolescents; Sleep; Actigraphy; Psychiatric Health
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents: Adolescents, male or female, ages 11 - 17. Participants will complete 7 days/nights of actigraphy and sleep-based EEG and questionnaires.

SUMMARY:
The overall goal of this study is to investigate associations between sleep/circadian disturbances and psychiatric health among adolescents recruited from primary and specialty health clinics.

DETAILED DESCRIPTION:
This project will involve recruitment of 100 adolescents from primary and specialty health clinics. Participants will participate in 3 phases: screening/intake visit, sleep study, and follow-up visit.

The 1-hour screening/intake visit will be conducted at the Duke ADHD clinic at 2608 Erwin Road, Pavilion East, Suite 300, Durham, NC 27705. During the screening/intake visit, participants and their parents will complete questionnaires regarding the adolescent's psychiatric health. Participants' vitals (i.e., height, weight, resting heart rate, blood pressure) will also be assessed and recorded.

Eligible participants will enter the 7-day sleep study, during which they will be asked to wear an actigraph watch 24 hours/day, apply a EEG sleep recorder each night, and complete a daily sleep diary.

Following the final night of the sleep study, participants and parents will be asked to return for a follow-up visit and will complete questionnaires about the participants' sleep over the past week.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Between the ages of 11 years 0 months to 17 years 11 months (inclusive), at the time of parental informed consent.
3. Ability to follow written and verbal instructions (English), as assessed by the PI and/or study coordinator.
4. Ability to comply with all testing, requirements, study procedures, and availability for the duration of the study.

Exclusion Criteria:

1. Participants who have a diagnosis of occult sleep disorders (i.e., sleep apnea, periodic leg movement syndrome)
2. Participants who currently use prescribed or over-the-counter sleep aids (i.e., melatonin)
3. Participants who have acute or chronic medical illnesses or medications that may interfere with sleep as determined by the research team.
4. Unable to comply with study requirements or otherwise unsuitable for participation in the opinion of the principal investigator.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents will be recruited from primary and specialty health clinics.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Psychiatric Health - Internalizing and Externalizing Symptoms of Childhood | 1 Day
  "Internalizing symptoms" and "Externalizing symptoms" subscales of the Child Behavior Checklist (CBCL)

SECONDARY OUTCOMES:
Acceptability of Devices - Tolerability Scale | 1 day
  Tolerability will be assessed using the At Home PSG Tolerability Scale, developed by Dr. Lunsford-Avery (PI) and colleagues. This scale measures comfort of devices while asleep and awake, sleep disturbances resulting from device use, and satisfaction with the devices.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Lunsford-Avery, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Child and Family Study Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lunsford-Avery JR, Keller C, Kollins SH, Krystal AD, Jackson L, Engelhard MM. Feasibility and Acceptability of Wearable Sleep Electroencephalogram Device Use in Adolescents: Observational Study. JMIR Mhealth Uhealth. 2020 Oct 1;8(10):e20590. doi: 10.2196/20590. PMID 33001035